CLINICAL TRIAL: NCT07069153
Title: Efficacy of Laser Therapy and Ozone Therapy for the Treatment of Oral Mucositis in Cancer Patients: A Randomized Clinical Trial
Brief Title: Laser vs Ozone Therapy for Oral Mucositis in Cancer Patients
Acronym: LOMUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-LOMUC
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Oral Mucositis; Head and Neck Neoplasms; Hematologic Neoplasms
Keywords: Oral Mucositis; Cancer Pain; Laser Therapy; Ozone Therapy; Photobiomodulation; Head and Neck Cancer; Hematologic Malignancies; Chemotherapy; Radiotherapy; Supportive Care in Oncology
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Hematologic Neoplasms; Cancer Pain | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Therapy for Oral Mucositis (Experimental): Patients in this arm will undergo high-power diode laser therapy using the Garda Laser LEO PLUS device with a flat-top handpiece at a wavelength of 660 nm. The laser is applied intraorally on the mucosal lesions following a standardized photobiomodulation protocol. The treatment is administered once daily for five consecutive days. Mucositis severity (WHO scale), pain intensity (VAS), and quality of life (OMWQ-HN) will be monitored from baseline through 30 days of follow-up.
  Interventions: Device: Laser Therapy
- Ozone Therapy for Oral Mucositis (Active Comparator): Patients in this arm will receive medical ozone therapy for the treatment of chemotherapy- or radiotherapy-induced oral mucositis. Ozone is administered intraorally in gaseous form using a Sweden & Martina DTA device and a flat probe specifically designed for mucosal application. The treatment is delivered once daily for five consecutive days, following a standardized therapeutic protocol. Clinical parameters including mucositis severity (WHO scale), pain (VAS), and quality of life (OMWQ-HN) will be assessed at baseline and during follow-up.
  Interventions: Device: Ozone therapy

INTERVENTIONS:
Device: Laser Therapy — High-power diode laser therapy is applied to the oral mucosa using the Garda Laser LEO PLUS device with a flat-top handpiece at 660 nm wavelength. Treatment is delivered once daily over five consecutive days according to a standardized photobiomodulation protocol (energy density: 2-4 J/cm²).
  Arms: Laser Therapy for Oral Mucositis
Device: Ozone therapy — Medical ozone gas is delivered intraorally using the Sweden & Martina DTA device. The treatment is administered once daily over five consecutive days. A flat-tipped probe is used to apply ozone directly to the mucosal lesions at a concentration of 30-40 µg/mL, following a standardized safety protocol.
  Arms: Ozone Therapy for Oral Mucositis

SUMMARY:
This randomized clinical trial aims to compare the efficacy of laser therapy and ozone therapy in the treatment of oral mucositis in adult cancer patients undergoing chemotherapy or radiotherapy, particularly those with head and neck tumors or hematologic malignancies. Oral mucositis is a frequent and debilitating complication of cancer treatment, characterized by painful ulcerations that impair nutrition, speech, and oral hygiene, often requiring opioid analgesics and supportive care.

Forty eligible patients will be randomly assigned to two parallel groups. The trial group will receive high-power diode laser therapy using a flat-top handpiece at 660 nm wavelength, following a standardized photobiomodulation protocol. The control group will be treated with medical ozone gas administered via an intraoral device, using a standardized ozone therapy protocol. Both treatments will be applied once daily over five consecutive days. Patients will be followed up at 15 and 30 days after treatment initiation.

The primary outcome is the reduction in mucositis severity, measured using the World Health Organization (WHO) Oral Toxicity Scale. Secondary outcomes include pain intensity assessed with the Visual Analogue Scale (VAS), and quality of life evaluated through the Oral Mucositis Weekly Questionnaire - Head and Neck (OMWQ-HN). The study seeks to determine whether laser therapy offers superior clinical benefits compared to ozone therapy in reducing lesion severity, alleviating pain, and improving patient well-being during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of head and neck cancer or hematologic malignancy
* Currently undergoing chemotherapy and/or radiotherapy
* Presence of oral mucositis of grade 2 or higher (WHO Oral Mucositis Scale)
* Ability to provide written informed consent
* Willingness to comply with study procedures and follow-up schedule

Exclusion Criteria:

* Presence of autoimmune or systemic diseases affecting the oral mucosa (e.g., lichen planus, pemphigus, pemphigoid)
* Presence of active oral infections unrelated to mucositis (e.g., candidiasis, herpes simplex)
* Previous treatment with ozone or laser therapy for oral mucositis in the past 3 months
* Pregnancy or breastfeeding
* Cognitive impairment or psychiatric disorders preventing full cooperation
* Known allergy or intolerance to ozone or laser exposure
* Use of investigational drugs or participation in other clinical trials within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Oral Mucositis Severity Assessed by WHO Oral Mucositis Scale | Baseline (T0), Day 5 (T1), Day 15 (T3), and Day 30 (T5)
  Oral mucositis severity will be evaluated using the World Health Organization (WHO) Oral Mucositis Scale, a standardized clinical tool that grades mucosal toxicity on a scale from 0 to 4. Grade 0 indicates no mucositis, grade 1 indicates soreness and erythema, grade 2 denotes erythema and ulcers but the patient can eat solid food, grade 3 represents ulcers with a liquid diet only, and grade 4 corresponds to severe mucositis with alimentation not possible. Scores will be recorded at baseline (T0), after 5 days of treatment (T1), and at follow-up visits on day 15 (T3) and day 30 (T5). The primary endpoint is the change in WHO score from baseline to day 30.

SECONDARY OUTCOMES:
Change in Pain Intensity Assessed by Visual Analogue Scale (VAS) | Baseline (T0), Day 5 (T1), Day 15 (T3), and Day 30 (T5)
  Pain intensity will be assessed using a 10 cm Visual Analogue Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain." Patients will be instructed to mark the point that best represents their current level of oral pain. VAS scores will be collected at baseline (T0), after each treatment session (T1-T5), and at follow-up visits on day 15 (T3) and day 30 (T5).
Change in Quality of Life Assessed by Oral Mucositis Weekly Questionnaire - Head and Neck (OMWQ-HN) | Baseline (T0), Day 5 (T1), Day 15 (T3), and Day 30 (T5)
  Quality of life will be assessed using the validated Oral Mucositis Weekly Questionnaire - Head and Neck (OMWQ-HN), a patient-reported outcome tool developed for individuals receiving radiotherapy or chemotherapy for head and neck cancer. The questionnaire includes 13 items covering oral pain, swallowing, speaking, eating, use of medications, and impact on daily life. Each item is scored on a 0 to 4 Likert scale, where 0 = "Not at all" and 4 = "Extremely." The overall OMWQ-HN score is calculated by summing all item scores, with total values ranging from 0 to 52. Higher scores indicate a greater negative impact on quality of life due to oral mucositis. The questionnaire will be administered at baseline (T0) and at day 30 (T5), allowing comparison of quality of life before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.